CLINICAL TRIAL: NCT00756106
Title: Quantitative Assessment of the Early and Late Effects of Radiation and Chemotherapy on Glioblastoma Using Multiple MRI Techniques
Brief Title: MRI Scans in Evaluating the Effects of Radiation Therapy and Chemotherapy in Patients With Newly Diagnosed Glioblastoma Multiforme or Anaplastic Glioma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding ended
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Elizabeth R. Gerstner, MD, MD, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 07-292
Record Dates: First submitted 2008-09-18; First posted 2008-09-19 (Estimated); Results first posted 2020-04-21 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-04

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult glioblastoma; adult giant cell glioblastoma; adult gliosarcoma; adult anaplastic astrocytoma; adult anaplastic ependymoma; adult anaplastic oligodendroglioma; adult mixed glioma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Gliosarcoma; Astrocytoma; Ependymoma; Oligodendroglioma; Glioma | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Temozolomide and Radiation Therapy (Experimental)
  Interventions: Drug: temozolomide; Other: Imaging biomarker analysis; Radiation: Photon Radiation Therapy

INTERVENTIONS:
Drug: temozolomide — Temozolomide is administered according to standard of care practice guidelines. Dosing may be modified at the discretion of the treating investigator.
Other: Imaging biomarker analysis — MRI
Radiation: Photon Radiation Therapy — Radiation is administered to the tumor plus edema with a 1-2 centimeter margin for a total dose of 60 Gy in 30 fractions.

SUMMARY:
RATIONALE: Diagnostic procedures, such as MRI, may help in learning how well radiation therapy and chemotherapy work in killing tumor cells and allow doctors to plan better treatment.

PURPOSE: This clinical trial is studying MRI scans to see how well they evaluate the effects of radiation therapy and chemotherapy in patients with newly diagnosed glioblastoma multiforme or anaplastic glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To quantitatively compare the relative cerebral blood volume/flow, mean transit time, and mean vessel diameter as measured by perfusion-weighted MRI before, during, and after chemoradiotherapy in patients with newly diagnosed glioblastoma multiforme.
* To measure the permeability-surface area product on a voxel-by-voxel basis before, during, and after chemoradiotherapy in these patients.
* To measure the full water self-diffusion tensor on a voxel-by-voxel basis before, during, and after chemoradiotherapy in these patients.
* To compare the tensor fractional anisotropy before, during, and after chemoradiotherapy in these patients.
* To compare the relative regional concentrations of choline, N-acetyl-asparate, and myoinositol as measured by magnetic resonance spectroscopy before, during, and after chemoradiotherapy to interrogate cell membrane turnover, neuronal integrity, and glial reactions.
* To test the affects of a short period of 100% oxygen inhalation on imaging of tumor and surrounding tissue regions of interest, specifically cerebral blood volume changes in each area as compared to room air.

Secondary

* To collect blood and urine samples for correlation analysis between imaging changes, molecular markers (including genetic markers), and clinical outcome of glioblastoma multiforme (phenotypic information).
* To correlate blood and urine biomarkers and blood genetic markers with tumor expression of these markers.

OUTLINE: Patients undergo radiotherapy once daily 5 days a week for 6 weeks. Patients also receive oral temozolomide once daily 7 days a week during radiotherapy. After completion of chemoradiotherapy, patients receive oral temozolomide once daily for 5 days. Treatment with temozolomide repeats every 28 days in the absence of disease progression or unacceptable toxicity.

Patients undergo MRI, including perfusion- and diffusion-weighted MRI, diffusion tensor imaging, and magnetic resonance spectroscopy prior to initiation of chemoradiotherapy, once weekly during chemoradiotherapy, and then monthly until tumor progression or until completion of 6 courses of post chemoradiotherapy.

After completion of study treatment, patients are followed annually.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly diagnosed anaplastic glioma (WHO grade III) or glioblastoma multiforme (WHO grade IV)
* Measurable disease

  * Residual tumor size after surgery ≥ 1 cm in one dimension
* Planning to undergo standard chemoradiotherapy with temozolomide

PATIENT CHARACTERISTICS:

* Glomerular filtration rate ≥ 60 mL/min
* Mini Mental Status Exam score > 15
* Sufficiently competent to give informed consent
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception during and for 2 months after completion of study treatment
* No contraindication to MRI or to use of the contrast agent gadolinium, including any of the following:

  * Claustrophobia
  * Metallic objects or implanted medical devices (e.g., cardiac pacemaker, aneurysm clips, surgical clips, prostheses, artificial hearts, valves with steel parts, metal fragments, shrapnel, tattoos near the eye, or steel implants)
  * Sickle cell disease
  * Renal failure
  * High risk for kidney disease (e.g., age > 60 years, diabetes, or history of systemic lupus erythematosus or multiple myeloma)
* No known history of chronic obstructive pulmonary disease or emphysema
* No other co-existing condition that, in the judgement of the investigator, may increase risk to the patient

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Non-VEGF investigational agent allowed
* No concurrent chemotherapy (other than temozolomide)
* No concurrent electron, proton, particle, or implant radiotherapy
* No concurrent stereotactic radiosurgery
* No concurrent anti-VEGF anti-tumor agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-07; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Gerstner, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hoebel KV, Bridge CP, Ahmed S, Akintola O, Chung C, Huang RY, Johnson JM, Kim A, Ly KI, Chang K, Patel J, Pinho M, Batchelor TT, Rosen BR, Gerstner ER, Kalpathy-Cramer J. Expert-centered Evaluation of Deep Learning Algorithms for Brain Tumor Segmentation. Radiol Artif Intell. 2024 Jan;6(1):e220231. doi: 10.1148/ryai.220231. PMID 38197800
- [Derived] Hoebel KV, Patel JB, Beers AL, Chang K, Singh P, Brown JM, Pinho MC, Batchelor TT, Gerstner ER, Rosen BR, Kalpathy-Cramer J. Radiomics Repeatability Pitfalls in a Scan-Rescan MRI Study of Glioblastoma. Radiol Artif Intell. 2020 Dec 16;3(1):e190199. doi: 10.1148/ryai.2020190199. eCollection 2021 Jan. PMID 33842889
- [Derived] Emblem KE, Farrar CT, Gerstner ER, Batchelor TT, Borra RJ, Rosen BR, Sorensen AG, Jain RK. Vessel caliber--a potential MRI biomarker of tumour response in clinical trials. Nat Rev Clin Oncol. 2014 Oct;11(10):566-84. doi: 10.1038/nrclinonc.2014.126. Epub 2014 Aug 12. PMID 25113840
- [Derived] Pinho MC, Polaskova P, Kalpathy-Cramer J, Jennings D, Emblem KE, Jain RK, Rosen BR, Wen PY, Sorensen AG, Batchelor TT, Gerstner ER. Low incidence of pseudoprogression by imaging in newly diagnosed glioblastoma patients treated with cediranib in combination with chemoradiation. Oncologist. 2014 Jan;19(1):75-81. doi: 10.1634/theoncologist.2013-0101. Epub 2013 Dec 5. PMID 24309981

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Temozolomide and Radiation Therapy
Started | 15
Completed | 3
Not Completed | 12

BASELINE CHARACTERISTICS:
Population: One participant withdrew consent after baseline and was excluded from the analysis set
Arm/Group | Temozolomide and Radiation Therapy
Number analyzed (Participants) | 14
Age, Continuous [Median (Full Range); unit: years] | 60 [35 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 14
Karnofsky Performance Status [Median (Full Range); unit: units on a scale] — The Karnofsky Performance Status is a measure of patients' general well-being and activities of daily living. The score ranges from 0 to 100, higher scores indicating a patient is better able to carry out daily activities.
  units on a scale | 90 [60 to 100]

OUTCOME MEASURES:

1. Primary Outcome: Relative Cerebral Blood Volume as Measured by Perfusion-weighted MRI Before, During, and After Chemoradiotherapy
Description: Relative cerebral blood volume (rCBV) is the blood volume in the region of interest (ROI) divided by the blood volume in the symmetrical region on the other side of the normal brain (control region). CBV was assessed using spin-echo post-contrast T1-weighted images. Multiple images were used to assess each participant at every time-point and the median value for each participant was calculated by time-point. The data presented represent the average of those median values at each time-point. The baseline value was measured twice (representing baseline 1 and 2) to make sure that the value was reproducible and to account for any variation attributable to measurement variation.
  CRT: Chemoradiotherapy Cx: The cycle number TMZ: temozolomide
Time Frame: Baseline, weekly during treatment, monthly following treatment for up to six months
Population: One participant withdrew consent after baseline and was excluded from the analysis set. The number of patients evaluated decreased over time due to participants experiencing disease progression and discontinuing from the study
Measure: Mean (Full Range); unit: ratio
Arm/Group | Temozolomide and Radiation Therapy
Number analyzed (Participants) | 14
ratio
  Baseline 1 | 0.88 [0.50 to 1.47]
  Baseline 2 | 0.90 [0.36 to 1.77]
  Week 1 CRT | 0.95 [0.47 to 1.78]
  Week 2 CRT | 1.0 [0.63 to 1.68]
  Week 3 CRT | 0.88 [0.39 to 1.58]
  Week 4 CRT | 0.83 [0.43 to 1.24]
  Week 5 CRT | 0.86 [0.43 to 1.33]
  Week 6 CRT | 0.76 [0.41 to 1.21]
  Pre-C1 TMZ | 0.68 [0.48 to 1.04]
  Pre-C2 TMZ: number analyzed (Participants) | 9
  Pre-C2 TMZ | 0.61 [0.45 to 0.83]
  Pre-C3 TMZ: number analyzed (Participants) | 8
  Pre-C3 TMZ | 0.59 [0.37 to 0.82]
  Pre-C4 TMZ: number analyzed (Participants) | 6
  Pre-C4 TMZ | 0.65 [0.38 to 0.87]
  Pre-C5 TMZ: number analyzed (Participants) | 5
  Pre-C5 TMZ | 0.61 [0.39 to 0.8]
  Pre-C6 TMZ: number analyzed (Participants) | 4
  Pre-C6 TMZ | 0.64 [0.18 to 1.30]
  Post-TMZ: number analyzed (Participants) | 3
  Post-TMZ | 0.32 [0.09 to 0.56]

2. Primary Outcome: Relative Cerebral Blood Flow as Measured by Perfusion-weighted MRI Before, During, and After Chemoradiotherapy
Description: Relative cerebral blood flow (rCBF) is the blood flow rate (the volume of blood passing through the specified are over a specified period of time) in the region of interest (ROI) divided by the blood flow rate in the symmetrical region on the other side of the normal brain (control region). CBF was assessed using spin-echo post-contrast T1-weighted images. CBF was assessed using spin-echo post-contrast T1-weighted images. Multiple images were used to assess each participant at every time-point and the median value for each participant was calculated by time-point. The data presented represent the average of those median values at each time-point. The baseline value was measured twice (representing baseline 1 and 2) to make sure that the value was reproducible and to account for any variation attributable to measurement variation.
  CRT: Chemoradiotherapy Cx: The cycle number TMZ: temozolomide
Time Frame: Baseline, weekly during treatment, monthly following treatment for up to six months
Population: as for outcome 1
Measure: Mean (Full Range); unit: ratio
Arm/Group | Temozolomide and Radiation Therapy
Number analyzed (Participants) | 14
ratio
  Baseline 1 | 0.83 [0.49 to 1.20]
  Baseline 2 | 0.86 [0.33 to 1.43]
  Week 1 CRT | 0.92 [0.59 to 1.37]
  Week 2 CRT | 0.94 [0.63 to 1.51]
  Week 3 CRT | 0.80 [0.46 to 1.38]
  Week 4 CRT | 0.79 [0.49 to 1.16]
  Week 5 CRT | 0.83 [0.48 to 1.30]
  Week 6 CRT | 0.73 [0.52 to 1.10]
  Pre-C1 TMZ | 0.63 [0.45 to 0.92]
  Pre-C2 TMZ: number analyzed (Participants) | 9
  Pre-C2 TMZ | 0.59 [0.5 to 0.69]
  Pre-C3 TMZ: number analyzed (Participants) | 8
  Pre-C3 TMZ | 0.60 [0.40 to 0.77]
  Pre-C4 TMZ: number analyzed (Participants) | 6
  Pre-C4 TMZ | 0.60 [0.52 to 0.67]
  Pre-C5 TMZ: number analyzed (Participants) | 5
  Pre-C5 TMZ | 0.52 [0.33 to 0.70]
  Pre-C6 TMZ: number analyzed (Participants) | 4
  Pre-C6 TMZ | 0.47 [0.30 to 0.66]
  Post-TMZ: number analyzed (Participants) | 3
  Post-TMZ | 0.37 [0.16 to 0.59]

3. Primary Outcome: Vessel Diameter as Measured by Perfusion-weighted MRI Before, During, and After Chemoradiotherapy
Time Frame: Baseline, weekly during treatment, monthly following treatment for up to six months
Population: Data not collected
Arm/Group | Temozolomide and Radiation Therapy
Number analyzed (Participants) | 0

4. Primary Outcome: Mean Transit Time as Measured by Perfusion-weighted MRI Before, During, and After Chemoradiotherapy
Description: Mean transit time (MTT) corresponds to the average time, in seconds, that red blood cells spend within a determinate volume of capillary circulation.
Time Frame: Baseline, weekly during treatment, monthly following treatment for up to six months
Population: Data not collected
Arm/Group | Temozolomide and Radiation Therapy
Number analyzed (Participants) | 0

5. Primary Outcome: Permeability-surface Area Product Before, During, and After Chemoradiotherapy
Description: Permeability-surface Area Product (Ktrans). Ktrans reflects the efflux rate of contrast from blood plasma into the tissue extravascular extracellular space (EES). Ktrans was assessed using post-contrast T1-weighted images. Multiple images were used to assess each participant at every time-point and the median value for each participant was calculated by time-point. The data presented represent the average of those median values at each time-point.
  CRT: Chemoradiotherapy Cx: The cycle number TMZ: temozolomide
Time Frame: Baseline, weekly during treatment, monthly following treatment for up to six months
Population: as for outcome 1
Measure: Mean (Full Range); unit: min ^-1
Arm/Group | Temozolomide and Radiation Therapy
Number analyzed (Participants) | 14
min ^-1
  Baseline 1 | 0.053 [0.015 to .138]
  Baseline 2 | 0.039 [0.012 to 0.075]
  Week 1 CRT | 0.055 [0.021 to 0.128]
  Week 2 CRT | 0.048 [0.018 to 0.105]
  Week 3 CRT | 0.055 [0.014 to 0.100]
  Week 4 CRT | 0.053 [0.010 to 0.107]
  Week 5 CRT | 0.058 [0.009 to 0.154]
  Week 6 CRT | 0.059 [0.016 to 0.127]
  Pre-C1 TMZ | 0.063 [0.012 to 0.152]
  Pre-C2 TMZ: number analyzed (Participants) | 9
  Pre-C2 TMZ | 0.042 [0.007 to 0.068]
  Pre-C3 TMZ: number analyzed (Participants) | 8
  Pre-C3 TMZ | 0.050 [0.025 to 0.106]
  Pre-C4 TMZ: number analyzed (Participants) | 6
  Pre-C4 TMZ | 0.058 [0.014 to 0.139]
  Pre-C5 TMZ: number analyzed (Participants) | 5
  Pre-C5 TMZ | 0.056 [0.004 to 0.137]
  Pre-C6 TMZ: number analyzed (Participants) | 4
  Pre-C6 TMZ | 0.060 [0.008 to 0.121]
  Post-TMZ: number analyzed (Participants) | 3
  Post-TMZ | 0.032 [0.010 to 0.054]

6. Primary Outcome: Apparent Diffusion Coefficient Before, During, and After Chemoradiotherapy
Description: Apparent diffusion coefficient (ADC) is a measure of the magnitude of diffusion (of water molecules) within tissue. ADC was assessed using post-contrast T1-weighted images. Multiple images were used to assess each participant at every time-point and the median value for each participant was calculated by time-point. The data presented represent the average of those median values at each time-point.
  CRT: Chemoradiotherapy Cx: The cycle number TMZ: temozolomide
Time Frame: Baseline, weekly during treatment, monthly following treatment for up to six months
Population: as for outcome 1
Measure: Mean (Full Range); unit: mm2/s
Arm/Group | Temozolomide and Radiation Therapy
Number analyzed (Participants) | 14
mm2/s
  Baseline 1 | 0.00110 [0.00078 to 0.00169]
  Baseline 2 | 0.00113 [0.00078 to 0.00209]
  Week 1 CRT | 0.00106 [0.00073 to 0.00145]
  Week 2 CRT | 0.00110 [0.00092 to 0.00136]
  Week 3 CRT | 0.00118 [0.00090 to 0.00156]
  Week 4 CRT | 0.00122 [0.00097 to 0.00154]
  Week 5 CRT | 0.00125 [0.00103 to 0.00158]
  Week 6 CRT | 0.00125 [0.00098 to 0.00154]
  Pre-C1 TMZ | 0.00132 [0.00107 to 0.00173]
  Pre-C2 TMZ: number analyzed (Participants) | 9
  Pre-C2 TMZ | 0.00127 [0.00101 to 0.00155]
  Pre-C3 TMZ: number analyzed (Participants) | 8
  Pre-C3 TMZ | 0.00108 [0.00043 to 0.00128]
  Pre-C4 TMZ: number analyzed (Participants) | 6
  Pre-C4 TMZ | 0.00133 [0.00112 to 0.00151]
  Pre-C5 TMZ: number analyzed (Participants) | 5
  Pre-C5 TMZ | 0.00148 [0.00069 to 0.00257]
  Pre-C6 TMZ: number analyzed (Participants) | 4
  Pre-C6 TMZ | 0.00179 [0.00140 to 0.00258]
  Post-TMZ: number analyzed (Participants) | 3
  Post-TMZ | 0.00140 [0.00005 to 0.00275]

7. Primary Outcome: Tensor Fractional Anisotropy Before, During, and After Chemoradiotherapy
Description: Fractional anisotropy (FA) is a measure of the directionality of the molecular motion of water.
Time Frame: Baseline, weekly during treatment, monthly following treatment for up to six months
Population: Data not collected
Arm/Group | Temozolomide and Radiation Therapy
Number analyzed (Participants) | 0

8. Primary Outcome: Relative Regional Concentrations of Choline, N-acetyl-asparate, and Myoinositol as Measured by Magnetic Resonance Spectroscopy Before, During, and After Chemoradiotherapy to Interrogate Cell Membrane Turnover, Neuronal Integrity, and Glial Reactions
Time Frame: Baseline, weekly during treatment, monthly following treatment for up to six months
Population: Data not collected
Arm/Group | Temozolomide and Radiation Therapy
Number analyzed (Participants) | 0

9. Primary Outcome: Affects of a Short Period of 100% Oxygen Inhalation on Imaging of Tumor and Surrounding Tissue Regions of Interest, Specifically Cerebral Blood Volume Changes in Each Area as Compared to Room Air
Time Frame: Baseline, weekly during treatment, monthly following treatment for up to six months
Population: Data not collected
Arm/Group | Temozolomide and Radiation Therapy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were not collected
Description: Adverse event data were not collected as a part of this study
Arm/Group | Temozolomide and Radiation Therapy
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes